CLINICAL TRIAL: NCT02730143
Title: Effect of High Altitude Exposure, Acclimatization and Re-exposure on Nocturnal Breathing Pattern in Lowlanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB15-2709_V1
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Effect of High Altitude
Keywords: Altitude; Nocturnal breathing pattern

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude exposure (Experimental): Acute high altitude exposure followed by 8 day acclimatization and re-exposure after 6 days at low altitude
  Interventions: Other: Altitude exposure

INTERVENTIONS:
Other: Altitude exposure — Altitude exposure

SUMMARY:
Prospective interventional trial in lowlanders evaluating the effect of acute exposure, acclimatization and re-exposure of high altitude on nocturnal breathing pattern.

DETAILED DESCRIPTION:
Respiratory polygraphies will be performed in Santiago de Chile, 520 m, over the course of 3 days. Participants will then travel by commercial airline (5 h flight) and by bus (3 h ride) to the ALMA base camp located at 2900 m near San Pedro de Atacama, northern Chile. Participants will stay there for the next 7 nights and respiratory polygraphies will be performed on night 1 and 6. They will be spend the days (6-8 h daily) at the telescope station at 5050 m while undergoing physiological testing. Daily transports from 2900 to 5050 m will be by car (1 h ride, one way). After the first 8 day altitude sojourn participants will return to the Santiago area (520 m) for a 6 day recovery period.

A second altitude sojourn with an identical schedule as the one described above and a final low altitude stay of 3 days will follow.

ELIGIBILITY:
Inclusion Criteria:

* born, raised and currently living <800m
* No overnight stay at altitudes >1500 m 4 weeks before the study

Exclusion Criteria:

* Previous altitude intolerance to altitude <3000 m
* Pregnancy
* Health impairment, which requires regular treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-05-07 (Actual); Study Completion 2016-05-07 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | first sojourn at 5050 m, night 1, 6; second sojourn at 5050 m, night 1, 6; low altitude sojourn at 520 m, night 1
  Change in mean nocturnal oxygen saturation over the course of high altitude exposure during 2 sojourns at 5050 m compared to low altitude

SECONDARY OUTCOMES:
Apnea-/hypopnea index measured by respiratory polygraphy | first sojourn at 5050 m, night 1, 6; second sojourn at 5050 m, night 1, 6; low altitude sojourn at 520 m, night 1
  Change in apnea-/hypopnea index over the course of high altitude exposure during 2 sojourns at 5050 m compared to low altitude
Oxygen desaturation index measured by respiratory polygraphy | first sojourn at 5050 m, night 1, 6; second sojourn at 5050 m, night 1, 6; low altitude sojourn at 520 m, night 1
  Change in oxygen desaturation index over the course of high altitude exposure during 2 sojourns at 5050 m compared to low altitude
Acute mountain sickness measured by the Environmental Symptom questionnaire cerebral score (AMSc) | first sojourn at 5050 m, day 2, 7; second sojourn at 5050 m, day 2,7; low altitude sojourn at 520 m, day 2
  Incidence of acute mountain sickness (AMSc score >= 0.7) over the course of high altitude exposure during 2 sojourns at 5050 m compared to low altitude

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waldner NF, Hartmann SE, Muralt L, Lichtblau M, Bader PR, Rawling JM, Lopez I, Ulrich S, Poulin MJ, Bloch KE, Furian M. Oxygen saturation and acute mountain sickness during repeated altitude exposures simulating high-altitude working schedules. Sci Rep. 2025 Apr 15;15(1):12987. doi: 10.1038/s41598-025-97554-7. PMID 40234589